CLINICAL TRIAL: NCT01980108
Title: Quantitative Ultrasound Assessment of Gastric Volume in Pregnant Women at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 13-07
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Respiratory Aspiration; Pregnancy
Keywords: Pregnancy; Respiratory Aspiration; Gastric Contents; Ultrasound
MeSH Terms: conditions — Respiratory Aspiration | interventions — Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- empty stomach (No Intervention): No fluid will be given to the patient prior to scanning.
- 50mL (Experimental): 50mL of water will be given to the patient prior to scanning
  Interventions: Other: water
- 100mL (Experimental): 100mL of water will be given to the patient prior to scanning
  Interventions: Other: water
- 200mL (Experimental): 200mL of water will be given to the patient prior to scanning
  Interventions: Other: water
- 300mL (Experimental): 300mL of water will be given to the patient prior to scanning
  Interventions: Other: water
- 400mL (Experimental): 400mL of water will be given to the patient prior to scanning
  Interventions: Other: water

INTERVENTIONS:
Other: water — water
  Arms: 100mL; 200mL; 300mL; 400mL; 50mL

SUMMARY:
Solid food or fluid residue in the stomach is always a major concern when patients need medical procedures under sedation or general anesthesia, due to the high risk of pulmonary aspiration of the stomach contents. This is especially important in emergency procedures, when a fasting period is not observed. The aspiration of the stomach contents into one's lungs can lead to serious complications (such as severe respiratory failure). Information from a bedside ultrasound assessment of the stomach may be a very useful tool to decide whether or not it's safe to proceed, cancel or delay a surgical procedure.

The investigotrs hypothesize that a mathematical model can be constructed to predict clear fluid volume in the stomach of non-labouring pregnant patients, as it has been developed in healthy adult volunteers.

DETAILED DESCRIPTION:
Food residue in the stomach of patients scheduled to have surgery is considered a major risk factor for pulmonary aspiration of gastric contents. The resulting respiratory compromise after aspiration is associated with significant morbidity and mortality. The risk of pulmonary aspiration is especially important in pregnant women, as they may often require surgery without having observed appropriate fasting. A bedside ultrasound assessment of the status of the gastric content would be of great value for the clinician. This technique has recently been shown very promising in non-pregnant patients and it is important to study its feasibility in the pregnant population.

In this study, patients fast overnight and are randomized to the following groups: empty, or various volumes of fluid (50, 100, 200, 300 or 400mL of apple juice before scanning). Their gastric contents are then assessed by an anesthesiologist, using ultrasound. The investigators aim to evaluate a standardized quantitative ultrasound assessment of gastric volume in non-labouring pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer non-labouring pregnant women at term (≥ 36 weeks)-
* 18 years or older
* ASA Physical Status I-III
* 50-120 kg of weight
* 150 cm of height or taller
* Ability to understand the rationale of the study assessments and to provide signed informed consent
* Written informed consent

Exclusion Criteria:

* Known pre-existing abnormal anatomy of the upper gastrointestinal tract
* History of upper GI tract surgical procedure

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Correlation between ingested volume and CSA in antrum | 5-10 minutes
  The patient will ingest 0, 50, 100, 200, 300 or 400mL of apple juice, and then the cross-sectional area (CSA) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Arzola, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada